CLINICAL TRIAL: NCT05930106
Title: Respiratory Variation of Carotid Doppler Peak Velocity in Liposuction Fluid Management
Brief Title: Carotid Doppler Peak Velocity Variation in Liposuction Fluid Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TJ Plast Advanced Center for Plastic Surgery (Other)
Responsible Party: Principal Investigator, Sergio Soto Hopkins, Principal Investigator, TJ Plast Advanced Center for Plastic Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2023-02
Record Dates: First submitted 2023-06-09; First posted 2023-07-05 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Lipodystrophy
Keywords: liposuction; carotid artery doppler peak velocity variation; plethysmography variability index; fluid ratio
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Intervention Model Description: The research will involve 50 female patients who have undergone liposuction and will be divided into two groups.
  Group Intraoperative Fluid Ratio: Fluid administration will be determined by the intraoperative fluid ratio. This ratio is calculated by dividing the sum of subcutaneous infiltration and intravenous fluid by the total aspirate volume. Depending on the aspiration volume, it will be maintained at 1-1.4.
  Group Carotid Artery Peak Velocity Variation: Patients will be given a fluid maintenance rate of 1.5 ml/kg/h. To determine fluid responsiveness, the carotid artery peak velocity variation (ΔVPeak-CA) will be measured before, during, and after the procedure. If the ΔVPeak-CA goes above 15%, the patient will receive a fluid bolus of lactated ringer solution at a rate of 4-6 ml/kg over 10-15 minutes, and the team will re-measure fluid responsiveness 10 minutes after each ΔVPeaK-CA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intraoperative fluid ratio (Active Comparator): The intraoperative fluid ratio will determine fluid administration. This ratio is calculated by dividing the sum of subcutaneous infiltration and intravenous fluid by the total aspirate volume. Depending on the aspiration volume, it will be maintained at 1-1.4.
  Interventions: Other: Intraoperative fluid ratio
- Group Carotid Artery Peak Velocity Variation (Experimental): Patients will be given a fluid maintenance rate of 1.5 ml/kg/h. To determine fluid responsiveness, the carotid artery peak velocity variation (ΔVPeak-CA) will be measured before, during, and after the procedure. If the ΔVPeak-CA goes above 15%, the patient will receive a fluid bolus of lactated ringer solution at a rate of 4-6 ml/kg over 10-15 minutes, and the team will re-measure fluid responsiveness 10 minutes after each ΔVPeaK-CA.
  Interventions: Device: Carotid Artery Doppler Peak Velocity Variation

INTERVENTIONS:
Other: Intraoperative fluid ratio — This ratio is calculated by dividing the sum of procedure subcutaneous infiltration and intravenous fluid by the total aspirate volume during surgery
  Arms: Group Intraoperative fluid ratio
Device: Carotid Artery Doppler Peak Velocity Variation — Patients will be given a fluid maintenance rate of 1.5 ml/kg/h. To determine fluid responsiveness, the carotid artery peak velocity variation (ΔVPeak-CA) will be measured before, during, and after the procedure. If the ΔVPeak-CA goes above 15%, the patient will receive a fluid bolus of lactated ringer solution at a rate of 4-6 ml/kg over 10-15 minutes, and the team will re-measure fluid responsiveness 10 minutes after each ΔVPeaK-CA.
  Arms: Group Carotid Artery Peak Velocity Variation

SUMMARY:
This study aims to compare the hemodynamic parameters, postoperative plethysmography variability index, the total amount of postoperative intravenous fluid administration needed, and the urine output of two methods of fluid resuscitation during liposuction surgery. One method involves using carotid artery Doppler peak velocity variation, while the other is the conventional fluid ratio.

DETAILED DESCRIPTION:
The research will involve 50 female participants who have undergone liposuction and will be divided into two groups.

Group 1: Fluid administration will be determined by the intraoperative fluid ratio. This ratio is calculated by dividing the sum of subcutaneous infiltration and intravenous fluid by the total aspirate volume. Depending on the aspiration volume, it will be maintained at 1-1.4.

Group 2: Participants will be given a fluid maintenance rate of 1.5 ml/kg/h. To determine fluid responsiveness, the carotid artery peak velocity variation (ΔVPeak-CA) will be measured before, during, and after the procedure. If the ΔVPeak-CA goes above 15%, the patient will receive a fluid bolus of lactated ringer solution at a rate of 4-6 ml/kg over 10-15 minutes, and the team will re-measure fluid responsiveness 10 minutes after each ΔVPeaK-CA.

During the examination, a single cardiothoracic anesthesiologist will use a 13-6 MHz linear probe (Fujifilm Sonosite M-Turbo) to measure the peak velocity of the carotid artery on the left side. The sample volume will be positioned at the center of the lumen, 2 cm from the bulb, and a pulsed wave Doppler examination will be conducted.

To measure the ΔVPeak-CA, the investigators will calculate the maximum and minimum values during one respiratory cycle. This will be done by using the formula: 100x (maximum peak velocity - minimum peak velocity) / [(maximum peak velocity + minimum peak velocity)/2].

Surgical technique

The superwet tumescence technique will be the only method utilized for infiltration during the procedure. All participants will undergo power-assisted liposuction, and a single surgeon will operate. The wetting solution will contain 1000cc of normal saline and 2mg of epinephrine in a 1:500,000 ratio. The total Infiltration volume will depend on the patient.

The total amount of aspiration will depend on the patient and surgery plan and can vary between 2500 to 5000 ml

During the surgical procedure, the investigators will monitor vital signs such as blood pressure, heart rate, temperature, oxygen levels, and urine output. Additionally, the investigators will track the amount of fluids given and removed, and the volume of blood aspirated.

Following surgery, participants will be hospitalized for 24 hours. During this time, the investigators will closely monitor the plethysmography variability index (PVI) in both groups. If the PVI exceeds 15%, participants will receive a ringer lactate fluid bolus of 4-6 ml/kg. Additionally, the investigators will keep track of their urine output, total fluid intake, and vital signs

ELIGIBILITY:
Inclusion Criteria:

* Female patients between 21 and 60 years old
* Liposuction with or without abdominoplasty
* American Society of Anesthesiologists Ӏ & ӀӀ.

Exclusion Criteria:

* History of previous liposuction surgery
* American Society of Anesthesiologist III
* Coagulation disorders
* Cardiopulmonary disorders

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Mean Postoperative PVi | 24 hours
  Following surgery, patients will be hospitalized for 24 hours. Throughout this period, the investigators will keep a close eye on the Plethysmography Variability Index (PVi) in both groups. The PVi is a dynamic index that measures the relative variability of the plethysmography waveform detected noninvasively from a pulse oximetry sensor, ranging from 0 to 100. By automatically calculating the dynamic changes that occur during the respiratory cycle, it uses the detected amplitudes. A higher variability in the plethysmography waveform has been linked to preload dependence and fluid responders. If the PVi exceeds 15%, the patient will receive a fluid bolus of lactated ringer solution at a rate of 4-6 ml/kg over 10-15 minutes.
Postoperative intravenous fluid balance | 24 hours
  Following surgery, patients will be hospitalized for 24 hours. During the postoperative period, the investigators will keep track and document the exact volume of fluid administered in milliliters.

SECONDARY OUTCOMES:
The intraoperative total volume of urine in the patient's catheter bag | the duration of the surgery
  During the intraoperative period, the investigators will measure and record the total volume of urine accumulated in the patient's catheter bag over the surgery period and will report urine output measured in milliliters per kilogram per hour.
The postoperative total volume of urine in the patient's catheter bag | 24 hours
  During the postoperative period, the investigators will measure and record the total volume of urine accumulated in the patient's catheter bag over a 24-hour period and will report urine output measured in milliliters per kilogram per hour.
Mean arterial blood pressure during hospitalization | 24 hours
  Following surgery, patients will be hospitalized for 24 hours. During this time, the investigators will monitor Mean arterial pressure
The intraoperative intravenous fluid balance | the duration of the surgery
  Throughout the surgical procedure, the investigators will meticulously monitor and record the precise amount of fluid administered in milliliters.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Soto Hopkins, M.D., Principal Investigator — TJ Plast Advanced Center for Plastic Surgery; Hector Milla, M.D., Study Chair — TJ Plast Advanced Center for Plastic Surgery; Israel Espino Gaucin, M.D., Study Director — TJ Plast Advanced Center for Plastic Surgery
Locations (1):
- TJ Plast out patient, S.A. de C.V., Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers interested in liposuction fluid management. Data will be coded, and approval consent forms it's a prerequisite.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 months after publication and for 24 months
Access Criteria: Qualified researchers can request access to IPD, and will be provided following the review and approval of the research proposal

REFERENCES:
- [Background] Wang G, Cao WG, Zhao TL. Fluid management in extensive liposuction: A retrospective review of 83 consecutive patients. Medicine (Baltimore). 2018 Oct;97(41):e12655. doi: 10.1097/MD.0000000000012655. PMID 30313055
- [Result] Song Y, Kwak YL, Song JW, Kim YJ, Shim JK. Respirophasic carotid artery peak velocity variation as a predictor of fluid responsiveness in mechanically ventilated patients with coronary artery disease. Br J Anaesth. 2014 Jul;113(1):61-6. doi: 10.1093/bja/aeu057. Epub 2014 Apr 9. PMID 24722322
- [Result] Ibarra-Estrada MA, Lopez-Pulgarin JA, Mijangos-Mendez JC, Diaz-Gomez JL, Aguirre-Avalos G. Respiratory variation in carotid peak systolic velocity predicts volume responsiveness in mechanically ventilated patients with septic shock: a prospective cohort study. Crit Ultrasound J. 2015 Dec;7(1):29. doi: 10.1186/s13089-015-0029-1. Epub 2015 Jun 26. PMID 26123610

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT05930106/Prot_SAP_ICF_000.pdf